CLINICAL TRIAL: NCT00748514
Title: Impact of a Capsular Incision on Biochemical Recurrence After Radical Perineal Prostatectomy
Brief Title: A Capsular Incision and Biochemical Recurrence After Radical Perineal Prostatectomy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Choi Han Yong, Samsung Medical Center,Sungkyunkwan University School of Medicine
Other Study IDs: SMC IRB 2008-08-012; SMC IRB 2008-08-012
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Radical Perineal Prostatectomy
Keywords: capsular incision; biochemical recurrence; radical perineal prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — prostate gland
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the impact of capsular incisions on biochemical recurrence (BCR) and the potential risk factors of capsular incisions.

DETAILED DESCRIPTION:
The pathological classification of the prostate following radical prostatectomy provides important prognostic information; an accurate pathology report is the cornerstone to cancer treatment and follow-up. In addition to the preoperative serum PSA, Gleason score on pathology specimens, seminal vesicle invasion and lymph node status, and a positive surgical margin with extraprostatic extension (EPE) are significant predictors of clinical and biochemical recurrence. However, the prognostic implication of a capsular incision, a tumor extending to the inked margins without a histologically documented EPE, remains to be defined.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven prostate cancer
* follow-up for at least 6 months

Exclusion Criteria:

* insufficient biopsy data
* seminal vesicle invasion or lymph node involvement on pathology
* neoadjuvant or adjuvant therapy

Ages: 43 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the prostate cancer patients treated with radical perineal prostatectomy at single tertiary institution
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 1995-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
biochemical recurrence of prostate cancer | upto the final date of study

SECONDARY OUTCOMES:
risk factors for capsular incisions | at surgery

CONTACTS AND LOCATIONS:
Overall Officials: han yong Choi, professor, Principal Investigator — Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Chuang AY, Nielsen ME, Hernandez DJ, Walsh PC, Epstein JI. The significance of positive surgical margin in areas of capsular incision in otherwise organ confined disease at radical prostatectomy. J Urol. 2007 Oct;178(4 Pt 1):1306-10. doi: 10.1016/j.juro.2007.05.159. Epub 2007 Aug 14. PMID 17698141
- [Result] Shuford MD, Cookson MS, Chang SS, Shintani AK, Tsiatis A, Smith JA Jr, Shappell SB. Adverse prognostic significance of capsular incision with radical retropubic prostatectomy. J Urol. 2004 Jul;172(1):119-23. doi: 10.1097/01.ju.0000132137.02846.ec. PMID 15201750